CLINICAL TRIAL: NCT01508013
Title: An Appearance-Based Intervention to Reduce Teen Skin Cancer Risk
Acronym: iSTART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, Joel Hillhouse, Professor, East Tennessee State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01CA134891-01A2 (NIH)
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-04

CONDITIONS: Skin Cancer
Keywords: Melanoma; Basal Cell Carcinoma; Squamous Cell Carcinoma
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Appearance-Focused Website Intervention (Experimental): This is a Internet-based appearance-focused prevention intervention based on the Behavioral Alternatives Model.
  Interventions: Behavioral: Appearance-Focused Website Intervention
- Control Website (Active Comparator): Control participants viewed an Internet site designed to provide drug and alcohol education for teens.
  Interventions: Behavioral: Control Website

INTERVENTIONS:
Behavioral: Appearance-Focused Website Intervention — The intervention is a teen-friendly website with information concerning the health and appearance effects of indoor tanning.
  Arms: Appearance-Focused Website Intervention
Behavioral: Control Website — The control website contains information about alcohol and drug abuse which is oriented for a teen audience.
  Arms: Control Website

SUMMARY:
The purpose of this study is to determine whether a skin cancer prevention website is effective at reduce female teenagers' desire to use indoor tanning and ultimately their use of indoor tanning over an 18 month period.

DETAILED DESCRIPTION:
The project is designed to improve the understanding of, and ability to affect UV risk behavior in teenage populations. The International Agency for Research in Cancer classifies indoor tanning as "carcinogenic to humans." There is evidence that female indoor tanning use increases dramatically from freshman to senior years of high school (e.g., 25-40% of older high school girls) making high school a critical time period for anti-tanning interventions to be carried out. This proposal assesses the effectiveness of a skin cancer prevention website for a nationally representative sample of high school teens in a randomized controlled trial. Teens exposed to the website will report reduced indoor tanning intentions, frequency and overall percentage of users while increasing sun protective behaviors at long-term (i.e 18 month) follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Teenager between 12 and 18 years old; has either indoor tanned in the past year or has indicated their intentions to indoor tan in the coming year.

Exclusion Criteria:

* None other than not meeting inclusion criteria.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 443 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel J Hillhouse, Ph.D., Principal Investigator — East Tennessee State University
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from high school teenage women who indoor tan. The final dataset will include self-reported demographic, attitudinal, cognitive and behavioral data from surveys about private personal behaviors. The final dataset will be stripped of identifiers prior to release for sharing. We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and to not attempting to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Groups:
- Appearance-Focused Website Intervention: This is a Internet-based appearance-focused prevention intervention based on the Behavioral Alternatives Model. Appearance-Focused Website Intervention: The intervention is a teen-friendly website with information concerning the health and appearance effects of indoor tanning.
- Control Website: Control participants viewed an Internet site designed to provide drug and alcohol education for teens. Control Website: The control website contains information about alcohol and drug abuse which is oriented for a teen audience.
Period: Overall Study
Arm/Group | Appearance-Focused Website Intervention | Control Website
Started | 214 | 229
Completed | 182 | 206
Not Completed | 32 | 23

BASELINE CHARACTERISTICS:
Population: Adolescent females aged 12-18 years old who expressed interest in future indoor tanning.
Groups:
- Total: Total of all reporting groups
Arm/Group | Appearance-Focused Website Intervention | Control Website | Total
Number analyzed (Participants) | 214 | 229 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.19 (1.89) | 15.24 (1.91) | 15.21 (1.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 229 | 443
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 28 | 54
  Not Hispanic or Latino | 188 | 201 | 389
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 214 | 229 | 443
Indoor Tanning Frequency [Mean (Standard Deviation); unit: Indoor tanning sessions] | 6.36 (25.29) | 5.94 (23.01) | 6.14 (24.11)
Indoor Tanning Intentions Scale [Mean (Standard Deviation); unit: units on a scale] — The Indoor Tanning Intentions Scale can range from 1 (definitely do not intend; better) to 7 (definitely do intend; worse).
  units on a scale | 4.14 (2.00) | 3.74 (2.01) | 3.93 (2.01)
Indoor Tanning Willingness Scale [Mean (Standard Deviation); unit: units on a scale] — The Indoor Tanning Willingness scale ranges from 1 (definitely not willing; better ) to 7 (definitely willing; worse).
  units on a scale | 4.66 (1.92) | 4.55 (1.85) | 4.60 (1.88)
Indoor Tanning Attitudes Scale [Mean (Standard Deviation); unit: units on a scale] — The Indoor Tanning Attitudes Scale can range from 3 (strongly negative attitudes toward indoor tanning; better) to 15 (strongly positive attitudes toward indoor tanning; worse)
  units on a scale | 9.67 (3.35) | 9.34 (3.35) | 9.50 (3.35)
Indoor Tanning Social Approval Scale [Mean (Standard Deviation); unit: units on a scale] — The Indoor Tanning Social Approval Scale can range from 3 (strong beliefs peers do not approve indoor tanning; better) to 15 (strong beliefs peers do approve indoor tanning; worse)
  units on a scale | 11.99 (2.54) | 11.23 (2.87) | 11.59 (2.74)
Indoor Tanning Skin Damage Susceptibility Scale [Mean (Standard Deviation); unit: units on a scale] — The Indoor Tanning Skin Damage Susceptibility scale can range from 5 (low perceived susceptibility to skin damage from indoor tanning; worse) to 25 (high perceived susceptibility to skin damage from indoor tanning; better).
  units on a scale | 18.79 (4.81) | 19.20 (4.61) | 19.00 (4.71)

OUTCOME MEASURES:

1. Primary Outcome: Indoor Tanning Behavior
Description: Self-report measure of the number of times the teenager has indoor tanned over 12 month time period. The self-report measure has been validated in previous studies.
Time Frame: 12 months
Population: Adolescent females aged 12-18 years old who expressed interest in indoor tanning in the future.
Measure: Mean (Standard Deviation); unit: Indoor tanning sessions over past year
Arm/Group | Appearance-Focused Website Intervention | Control Website
Number analyzed (Participants) | 182 | 206
Indoor tanning sessions over past year | 5.29 (14.89) | 6.30 (16.08)
Statistical Analysis 1: Comparison: Appearance-Focused Website Intervention vs Control Website; Test type: Superiority or Other; p = .633, Mixed Models Analysis

2. Primary Outcome: Indoor Tanning Intentions
Description: A validated measure of the teenagers intentions to use indoor tanning in the next 12 months. Indoor tanning intentions are measured on a scale that ranges from 1 (definitely do not intend to indoor tan; better) to 7 (definitely do intend to indoor tan; worse).
Time Frame: 12 months
Population: Adolescent females aged 12-18 years old who expressed interest in indoor tanning in the next year.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Appearance-Focused Website Intervention | Control Website
Number analyzed (Participants) | 182 | 206
units on a scale | 2.91 (1.96) | 3.28 (2.10)
Statistical Analysis 1: Comparison: Appearance-Focused Website Intervention vs Control Website; Test type: Superiority or Other; p = .001, Mixed Models Analysis

3. Primary Outcome: Indoor Tanning Willingness
Description: Scale that measures adolescents willingness to indoor tan in the future. Indoor tanning willingness is measured on a scale that ranges from 1 (definitely not willing; better) to 7 (definitely willing; worse).
Time Frame: 12 months
Population: Adolescent females aged 12-18 years old that expressed interest in indoor tanning in the future.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Appearance-Focused Website Intervention | Control Website
Number analyzed (Participants) | 182 | 206
units on a scale | 3.34 (2.16) | 3.73 (62.22)
Statistical Analysis 1: Comparison: Appearance-Focused Website Intervention vs Control Website; Test type: Superiority or Other; p = .018, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Appearance-Focused Website Intervention | Control Website
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/206
Other Adverse Events (participants affected / at risk) | 0/182 | 0/206

LIMITATIONS AND CAVEATS:
None noted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No